CLINICAL TRIAL: NCT07100041
Title: The Effect of Breathing Exercises and Stress Ball Use During Dressing Changes on Pain, Anxiety, Comfort and Vital Signs in Burn Patients
Brief Title: Use of Breathing Exercises and Stress Balls During Dressing Changes in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Senem Andı, Master of Science in Nursing, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKU-SBF-SA-02
Record Dates: First submitted 2025-07-22; First posted 2025-08-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Breathing Exercise; Burns (Physical Finding); Pain; Pain Management; Stress Ball
Keywords: anxiety; breathing exercise; burns; pain; pain management; stress ball
MeSH Terms: conditions — Anxiety Disorders; Burns; Pain; Agnosia | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The study consists of three groups: a control group, a breathing exercise group, and a stress ball group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Standard Treatment) Group (Experimental): The standard dressing procedure in the control group is as follows: The protective covering over the wound is removed, and the wound is washed with an irrigation solution. Appropriate medications (decontamination and moisturising gel, debridement gel, alginate, antibiotics, and medications that promote cell regeneration) are applied based on the condition of the wound. A non-adhesive wound care dressing is then placed over the wound, and gauze is applied on top to cover it. Analgesia is not routinely administered in standard wound care. The dressing procedure takes an average of 5 minutes, depending on the size of the burn wound. In the control group, before the dressing procedure, the patient who volunteered to participate in the study will be given a patient information form, a burn-specific pain anxiety scale, and the pain level before dressing will be recorded using the Visual Analogue Scale (VAS) and vital signs will be checked, after which the standard dressing procedure will be
  Interventions: Other: Control (Standard Treatment) Group
- Breathing Exercise Group (Experimental): Before the dressing procedure, patients who volunteer to participate in the study will be given a patient information form, a burn-specific pain anxiety scale, and their pain level before dressing will be recorded using the GAS. After their vital signs are checked, they will be given a practical demonstration of breathing exercises. The breathing exercise will first be explained verbally by the project coordinator in the burn centre's training room, followed by a practical demonstration. The patient will then be asked to perform the exercise. Once the project coordinator is confident that the patient has learned how to perform the breathing exercise, the patient will be taken to the dressing room. During the standard dressing procedure, the patient will be instructed to continue performing the breathing exercise. Immediately before the dressing change, the patient will be positioned comfortably, and they will be instructed to use the breathing exerci
  Interventions: Other: Breathing Exercise Group
- Stress Ball Group (Experimental): The stress ball is made of a medium-hard plastic material that can be easily held in the hand. Before the dressing procedure, patients who volunteer to participate in the study will be given information about the use of the stress ball after the patient information form, the burn-specific pain and anxiety scale, and the pain level before dressing have been recorded using the GAS, and their vital signs have been checked. During the standard dressing procedure, patients will be instructed to squeeze and release the stress ball periodically until the dressing procedure is complete, focusing solely on the stress ball during this time (Ozen et al., 2023) (Kasar et al., 2020). A separate stress ball will be used for each patient in the stress ball group to ensure that the effectiveness of the stress ball remains consistent. To support patients' relaxation during the dressing procedure, a stress ball usage guide prepared by the project team will be provided via tablet. The
  Interventions: Other: Stress Ball Group

INTERVENTIONS:
Other: Breathing Exercise Group — Before the dressing procedure, patients who volunteer to participate in the study will be given a patient information form, a burn-specific pain anxiety scale, and their pain level before dressing will be recorded using the GAS. After their vital signs are checked, they will be given a practical demonstration of breathing exercises. The breathing exercise will first be explained verbally by the project coordinator in the burn centre's training room, followed by a practical demonstration. The patient will then be asked to perform the exercise. Once the project coordinator is confident that the patient has learned how to perform the breathing exercise, the patient will be taken to the dressing room. During the standard dressing procedure, the patient will be instructed to continue performing the breathing exercise. Immediately before the dressing change, the patient will be positioned comfortably, and they will be instructed to use the breathing
  Arms: Breathing Exercise Group
Other: Stress Ball Group — The stress ball is made of a medium-hard plastic material that can be easily held in the hand. Before the dressing procedure, patients who volunteer to participate in the study will be given information about the use of the stress ball after the patient information form, the burn-specific pain and anxiety scale, and the pain level before dressing have been recorded using the GAS, and their vital signs have been checked. During the standard dressing procedure, patients will be instructed to squeeze and release the stress ball periodically until the dressing procedure is complete, focusing solely on the stress ball during this time (Ozen et al., 2023) (Kasar et al., 2020). A separate stress ball will be used for each patient in the stress ball group to ensure that the effectiveness of the stress ball remains consistent. To support patients' relaxation during the dressing procedure, a stress ball usage guide prepared by the project team will be provided
  Arms: Stress Ball Group
Other: Control (Standard Treatment) Group — The standard dressing procedure in the control group is as follows: The protective covering over the wound is removed, and the wound is washed with an irrigation solution. Appropriate medications (decontamination and moisturising gel, debridement gel, alginate, antibiotics, and medications that promote cell regeneration) are applied based on the condition of the wound. A non-adhesive wound care dressing is then placed over the wound, and gauze is applied on top to cover it. Analgesia is not routinely administered in standard wound care. The dressing procedure takes an average of 5 minutes, depending on the size of the burn wound. In the control group, before the dressing procedure, the patient who volunteered to participate in the study will be given a patient information form, a burn-specific pain anxiety scale, and the pain level before dressing will be recorded using the Visual Analogue Scale (VAS) and vital signs will be checked,
  Arms: Control (Standard Treatment) Group

SUMMARY:
In burn patients, failure to effectively manage pain and pain-related anxiety negatively affects the healing process; therefore, pain and anxiety must be carefully managed in burn patients. In addition to managing pain and anxiety, providing comfort-based care also contributes to improving the individual's health and recovery. In this study, the effect of breathing exercises and stress ball use during dressing changes on pain, anxiety, and vital signs in burn patients will be evaluated.

DETAILED DESCRIPTION:
Patients who visited the outpatient clinic providing services to ambulatory patients at the Burn Centre of Adana City Training and Research Hospital of the Ministry of Health of the Republic of Turkey during the study period will constitute the study population. The sample size calculation for the study was performed using the G-Power 3.1 computer program. While this study does not evaluate the effects of breathing exercises and stress balls on pain and anxiety during wound or burn dressing changes, there are studies in the literature that have evaluated the effectiveness of both methods during various invasive procedures. Considering that the stress ball and breathing exercise groups will be compared with the control group in terms of pain and anxiety averages using t, and evaluating that the effect values in the studies in the literature vary between d=0.2 and d=0.8, According to Cohen, d=0.5, with 80% power at a 95% confidence interval, the total sample size is estimated to be 196 patients, with 64 patients in each group. Considering a 10% loss rate among patients, 70 patients will be included in each group at the beginning of the study, resulting in a total of 210 patients.

Participants who meet the inclusion criteria and volunteer will be provided with information about the study, and their verbal and written consent will be obtained. Prior to the dressing procedure, the patient information form will be completed, pain levels will be recorded using the Visual Analogue Scale (VAS), vital signs will be checked, and the Burn-Specific Pain Anxiety Scale (BSPAS) will be administered. Then, the GAS will be used to assess the pain level during the dressing procedure, and the pain level will be recorded. After the dressing, vital signs will be re-checked as soon as possible, and the General Comfort Scale Short Form (GCS-SF) will be administered. Data will be collected using the same data collection tools during the patient's two consecutive dressing changes (patients' dressings are changed every two days).

Block randomisation will be used to determine the groups in the study. Participants will be assigned to groups at the time of their outpatient visit, after eligibility criteria have been assessed. The homogeneity of the groups will be determined using a web-based randomisation system, Research Randomizer (https://www.randomizer.org/). A block randomisation list will be obtained for the three groups. Patients will be assigned to the intervention groups according to the obtained randomisation list.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65, seeking outpatient treatment at the burn centre,
* Without mental, hearing, visual or physical disabilities,
* Able to speak and understand Turkish,
* With a burn injury of 15% or less of the total body surface area (TBSA) and requiring dressing changes,
* At least three days have passed since the burn injury (the wound has passed the inflammatory phase of healing),
* Not in the maturation phase of wound healing,
* Burn area is on the hand, arm, leg, foot, or torso,
* No active burns on the hands,
* No respiratory issues.

Exclusion Criteria:

* Patients with neurological or psychiatric disorders,
* Patients with burns covering less than 15% of their body surface area or with no second-degree burns,
* Patients with burns in areas other than the hands, arms, legs, feet, and torso,
* Patients admitted to the burn centre,
* Patients with inhalation burns,
* Patients who receive sedation during dressing changes,
* Patients with complications such as infection or bleeding in the burn area,
* Patients who use pharmacological or non-pharmacological methods that may affect pain during dressing changes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Results | immediately before dressing, during dressing, immediately after dressing
  The VAS is a 10 cm horizontal line with numbers from 0 to 10, representing no pain at the start and the most severe pain that patients can feel at the end. On the scale, "0" means no pain and "10" means very severe pain. Participants are asked to select a number between "0" and "10" according to the degree of pain they feel.

SECONDARY OUTCOMES:
Patient Identification and Demographic Information Form | 5 minutes before the first dressing change
  The patient information form was created by the researcher based on relevant literature and consists of a total of 13 questions, including 8 questions related to demographic information and 5 questions related to burns.
Burn-Specific Pain Anxiety Scores Assessed Before Dressing | immediately before dressing
  Burn-Specific Pain Anxiety scale was developed by Taal and Faber in 1997 and measures the expected pain anxiety in burn patients during painful procedures such as dressing changes (Taal & Faber, 1997). The validity and reliability of the scale in Turkish were established by Deniz Doğan and Arslan (Deniz Doğan & Arslan, 2019). The scale consists of a total of eight items and is scored on a scale of 0 ('not at all') to 10 ('as badly as possible'). The lowest possible score is 0 and the highest possible score is 80. An increase in the score indicates an increase in the patient's anxiety due to painful procedures during their hospital stay. In the study conducted by Deniz Doğan and Arslan, the Cronbach's alpha coefficient was found to be 0.95 (Deniz Doğan & Arslan, 2019).
Patient Comfort Measured After Wound Dressing | immediately after dressing
  The General Comfort Scale Short Form was developed by Kolcaba and colleagues, and its validity and reliability in Turkish were established by Sarıtaş and colleagues (Kolcaba, Tilton, et al., 2006), (Sarıtaş et al., 2018). The scale is a six-point Likert type scale consisting of 28 items. The subscales of the scale are relief (items 1-9), relaxation (items 10-18), and superiority (items 19-28), and the items on the scale are scored between 28 and 168. The negative items in the scale are reverse-coded and summed. The total score is divided by the total number of scale items to find the mean score. In Sarıtaş and colleagues' study, the Cronbach's alpha coefficient of the scale was found to be 0.82 (Sarıtaş et al., 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health Adana City Training and Research Hospital Burn Centre, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to protect ethical constraints and participant confidentiality.

REFERENCES:
- [Background] Sarıtaş, S. Ç., Çevik, S., & Özden, G. (2018). Genel Konfor Ölçeği Kısa Formunun Türkçe Geçerlik ve Güvenirlik Çalışlması. Diyabet, Obezite ve Hipertansiyonda Hemflirelik Forumu Dergisi, 10(2), 16-22.
- [Background] Kolcaba K, Tilton C, Drouin C. Comfort Theory: a unifying framework to enhance the practice environment. J Nurs Adm. 2006 Nov;36(11):538-44. doi: 10.1097/00005110-200611000-00010. PMID 17099440
- [Background] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973
- [Background] Aktas GK, Ilgin VE. The Effect of Deep Breathing Exercise and 4-7-8 Breathing Techniques Applied to Patients After Bariatric Surgery on Anxiety and Quality of Life. Obes Surg. 2023 Mar;33(3):920-929. doi: 10.1007/s11695-022-06405-1. Epub 2022 Dec 8. PMID 36480101
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Fatma Eti Aslan. (2004). Sensitivity and selectivity of visual analog scale and the verbal rating scale in the assessment of postoperative pain. J. Intensive Care Nurs., 8, 1-6.
- [Background] 4. Bozorgnejad, M., Zarei, M. R., Mamashli, L., & Mohaddes Ardebili, F. (2019). The Effect of Rhythmic Breathing on the Anxiety of Dressing Change in Burning Patients. International Electronic Journal of Medicine, 8(2), 95-100. https://doi.org/10.34172/iejm.2019.04
- [Background] Najafi Ghezeljeh T, Mohades Ardebili F, Rafii F. The effects of massage and music on pain, anxiety and relaxation in burn patients: Randomized controlled clinical trial. Burns. 2017 Aug;43(5):1034-1043. doi: 10.1016/j.burns.2017.01.011. Epub 2017 Feb 4. PMID 28169080
- [Background] 7. Erbay, Ö., Yıldırım, Y., Fadıloğlu, Ç., & Şenuzun Aykar, F. (2019). Use of the Kolcaba's Comfort Theory in the Nursing Management of a Case with a Colostomy Opened Due to Rectum Cancer. Journal of Traditional Medical Complementary Therapies, 2(1), 42-48. https://doi.org/10.5336/jtracom.2019-64998
- [Background] Lee HW, Ang L, Kim JT, Lee MS. Aromatherapy for Symptom Relief in Patients with Burn: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2021 Dec 21;58(1):1. doi: 10.3390/medicina58010001. PMID 35056310